CLINICAL TRIAL: NCT03589456
Title: Establishment of a Registry for Patients Treated With Photodynamic Therapy (PDT)
Brief Title: Establishment of a PDT Patient Registry
Status: Terminated | Type: Observational
Why Stopped: Study was closed to accrual on January 15, 2020.
Sponsor: Concordia Laboratories Inc. (Industry)
Collaborators: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CLI-PDT1801_I 69818
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Lung Cancer
Keywords: lung cancer; lung carcinoma; lung metastases; metastases
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — There are no interventions associated with this registry as it is purely observational.

SUMMARY:
This is a non-intervention patient registry to gather data on the use of photodynamic therapy under real-life conditions. It will involve up to 20 sites in USA.

DETAILED DESCRIPTION:
The purpose of this patient registry is to collect information about a patient's cancer treatment, photodynamic therapy (PDT), used alone or in combination with surgery, chemotherapy and radiotherapy. Patients will be registered either before or after PDT is performed, regardless of the indication. Analysis of this information may help to refine the treatment care. Data collected in the registry includes patient characteristics/demographics, disease characteristics, treatment details (photodynamic therapy, radiation, chemotherapy, surgery, etc.), side effects, and survival outcomes. By participating in this registry, patients will not be asked to do anything that would not ordinarily be done as a matter of routine care including clinical assessments, laboratory tests, radiology procedures, and treatments. Information on disease, condition, and treatment will be recorded in the registry during routine visits.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (≥ 18 years of age) treated with PDT.
* Women and men and members of all races and ethnic groups.
* Subjects may have received prior treatment for their cancer.
* Subjects to give a written informed consent for prospectively collected data.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: It is intended to enroll all types of subjects requiring PDT for cancer.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-01-18 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
PDT Outcome | Up to 5-year follow-up
  Collection of information on patient characteristics, disease sites, and utilization of prior or combined treatments to evaluate the impact of these parameters on the treatment outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Gollnick, Ph.D., Principal Investigator — Roswell Park Cancer Institute
Locations (10):
- United States (10):
  - John Muir Clinical Research Center, Concord, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - University of Chicago, Chicago, Illinois
  - Alexian Brothers Hospital Network, Lisle, Illinois
  - Duke University Medical Center, Durham, North Carolina
  - Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin